CLINICAL TRIAL: NCT02178904
Title: Dual Energy Computed Tomography for Ischemia Determination Compared to "Gold Standard" Non-Invasive and Invasive Techniques
Brief Title: Dual Energy CT for Ischemia Determination Compared to "Gold Standard" Non-Invasive and Invasive Techniques
Acronym: DECIDE-Gold
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1309014314; R01HL111141 (NIH)
Record Dates: First submitted 2014-06-24; First posted 2014-07-01 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Ischemia
Keywords: Ischemia; Dual Energy Computed Tomography; Computed Tomographic Perfusion; Fractional Flow Rate; Invasive Coronary Angiography; Coronary Artery Stenosis
MeSH Terms: conditions — Ischemia; Coronary Stenosis | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suspected Coronary Artery Disease: Subjects with symptoms suspicious of obstructive CAD who are referred for non-emergent clinically-indicated invasive coronary angiography or stress-rest MPI. Intervention: Procedure/Surgery: CT and stress test
  Interventions: Procedure: CT and stress test

INTERVENTIONS:
Procedure: CT and stress test — Coronary computed tomographic angiography (CCTA) plus computed tomography stress myocardial perfusion imaging (CTP)

SUMMARY:
The purpose of this study is determine the diagnostic performance of dual energy computed tomography perfusion for non-invasive assessment of the hemodynamic significance of coronary stenosis, as compared to a direct measurement of fraction flow reserve during cardiac catheterization as a reference standard.

The overall objective of the present study is to determine the diagnostic performance of dual energy computed tomography perfusion for non-invasive assessment of the hemodynamic significance of coronary stenosis, as compared to direct measurement of fraction flow reserve during cardiac catheterization as a reference standard.

DETAILED DESCRIPTION:
Coronary artery disease is the leading cause of morbidity and mortality in the United States. At present, professional guidelines endorse the use of an array of non-invasive tests for patients with suspected coronary artery disease, which are limited to one of two approaches: 1) physiologic demonstration of ischemia by functional stress testing or 2) anatomic visualization of stenosis by coronary computed tomographic angiography.

Stress test for physiologic assessment of coronary disease is performed most commonly with the prognostic value unsurpassed by other non-invasive tests, with risk of cardiac events escalating exponentially with increasing inducible hypoperfusion. However, despite its high reported performance, the "real world" accuracy of stress test is less sanguine and demonstrates generally poor discrimination of specific vessels that accommodate coronary lesions that cause ischemia. These findings have encouraged the adoption of other stress tests, such as positron emission tomography, which offers reliable attenuation correction, increased count sensitivity, lower radiation dose and enhanced diagnostic performance. Positron emission tomography also enables measures of absolute myocardial blood flow.

Coronary computed tomographic angiography is an alternative test that evaluates coronary disease by direct anatomic visualization of stenoses in a manner similar to cardiac catheterization. Similarly, when employing invasive fractional flow reserve to identify ischemia, high-grade stenoses observed by computed tomography are causal of ischemia less than half of the time.

Multicenter randomized trial data examining invasive methods have demonstrated that a combined anatomic-physiologic approach by catheterization with fractional flow reserve improves identification of patients who may benefit from revascularization, by restricting revascularization to those with high-grade stenoses that specifically cause ischemia. Nevertheless, the combination of catheterization with fractional flow reserve is invasive, is not widely adopted in clinical practice, and is costly.

Computed tomography perfusion is a novel non-invasive technique that can evaluate the physiologic significance of coronary disease, and is performed by adding a single image acquisition to computed tomography in the same setting. The combination of computed tomography perfusion to computed tomography may represent an ideal "one-stop shop" that may allow for both anatomic and physiologic evaluation of coronary disease, serve as a more effective gatekeeper to cardiac catheterization, and better identify patients that would benefit from revascularization.

The emergence of dual energy computed tomography techniques enables potentially improved perfusion assessment. In particular, projection-based dual energy computed tomography is a novel computed tomography method that incorporates energy-dependent models for basis material decomposition within tissue, and may allow for absolute quantification of myocardial blood [iodine] volume with high accuracy and allows for single energy monochromatic imaging that retains image stability while reducing common computed tomography artifacts. Both of these measures by projection-based dual energy computed tomography enable quantitative assessment of myocardial iodine uptake, but the diagnostic performance of dual energy computed tomography as compared to nuclear stress testing has not been tested systematically to date.

To date, an integrated anatomic-physiologic approach by non-invasive methods has been lacking, largely due to the lack of a test that is capable of providing both accurate anatomic and physiologic data in a single setting.

The DECIDE-Gold trial will be a prospective multicenter study to evaluate the diagnostic performance of the dual energy computed tomography perfusion for the detection and exclusion of hemodynamically significant coronary artery disease, as defined by fractional flow reserve, the reference standard. The targeted population is subjects with suspected coronary artery disease who are referred for non-emergent clinically-indicated invasive coronary angiography or rest-stress nuclear imaging. The study is considered non-significant risk as investigators will be blinded to the dual energy computed tomography perfusion analyses will in no part play a role in the subject's medical treatment or clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients provide written informed consent
* Patients scheduled to undergo clinically-indicated non-emergent invasive coronary angiography
* suspected coronary artery disease

Exclusion Criteria:

* Suspicion of acute coronary syndrome (acute myocardial infarction and unstable angina)
* Recent prior myocardial infarction within 40 days of ICA
* Known complex congenital heart disease
* Significant arrhythmia or tachycardia
* Impaired chronic renal function (serum creatinine > 1.5 mg/dl or GFR < 30 ml/min)
* Patients with known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status
* Contraindication to adenosine, including 2nd or 3rd degree heart block; sick sinus syndrome; long QT syndrome; severe hypotension, severe asthma, severe COPD or bronchodilator-dependent COPD
* Patient requires an emergent procedure
* Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, and severe congestive heart failure (NYHA III or IV) or acute pulmonary edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals in Argentina, Beijing, Seattle, Vancouver, New York
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of dual energy CCTA plus perfusion (DECTP) to determine presence or absence of at least one hemodynamically (HD)-significant coronary artery stenosis* at the subject-level when compared to FFR. | Within 60 days between CT and cath
  Diagnostic accuracy of coronary computed tomography angiography plus dual energy computed tomographic perfusion to determine presence or absence of at least one hemodynamically-significant coronary artery stenosis at the subject level when compared to fractional flow reserve as the reference standard.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value of coronary computed tomography angiography plus DECTP at the subject level using binary outcomes when compared to fractional flow reserve as the reference standard. | Within 60 days between tests
  Sensitivity, specificity, positive predictive value, and negative predictive value of coronary computed tomography angiography plus dual energy computed tomographic perfusion at the subject level using binary outcomes when compared to fractional flow reserve as the reference standard.
Diagnostic performance (accuracy, sensitivity, specificity, PPV, and NPV) of CCTA plus DECTP for HD-significant stenosis* at the vessel-level when compared to FFR. | Within 60 days between tests
  Diagnostic performance (sensitivity, specificity, positive predictive value, and negative predictive value) of coronary computed tomography angiography plus dual energy computed tomographic perfusion for the presence or absence of hemodynamically-significant coronary artery stenosis at the vessel level using binary outcomes when compared to fractional flow reserve as the reference standard.

OTHER OUTCOMES:
Diagnostic accuracy of DECTP alone for HD-significant stenosis* at the subject-level and vessel-level when compared to FFR. | Within 60 days between tests
  Diagnostic accuracy of dual energy computed tomographic perfusion alone to determine presence or absence of at least one hemodynamically-significant coronary artery stenosis at the subject level using binary outcomes when compared to fractional flow reserve as the reference standard.
Diagnostic accuracy of CCTA plus DECTP for HD-significant stenosis at the subject-level and vessel-level when compared to MPI. | Within 60 days between tests
  Sensitivity, specificity, positive predictive value, and negative predictive value of dual energy computed tomographic perfusion alone at the subject level using binary outcomes when compared to fractional flow reserve as reference standard.
Diagnostic accuracy of DECTP alone for HD-significant stenosis at the subject-level and vessel-level when compared to MPI. | Within 60 days between tests
  Diagnostic performance (accuracy, sensitivity, specificity, positive predictive value and negative predictive value) of dual energy computed tomographic perfusion alone for the presence or absence of hemodynamically-significant coronary artery stenosis at the vessel level using binary outcomes when compared to fractional flow reserve as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Leslee J Shaw, PhD, Principal Investigator — NewYork-Presbyterian Hospital and the Weill Cornell Medical College
Locations (5):
- United States (5):
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Weill Cornell Medical College, New York, New York
  - Wexner Medical Center, The Ohio State University Medical Center, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided